CLINICAL TRIAL: NCT04645953
Title: A Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of Staccato Granisetron (AZ-010) for the Acute Treatment of Moderate to Severe Cyclic Vomiting Syndrome
Brief Title: Staccato Granisetron® (AZ 010) for the Treatment of Cyclic Vomiting Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMDC 010-201
Record Dates: First submitted 2020-11-16; First posted 2020-11-27 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Cyclic Vomiting Syndrome
Keywords: Cyclic Vomiting Syndrome; CVS; Vomiting; Retching; Abdominal migraine; Nausea; Stomach pain; Unexplained vomiting; Functional GI Disorder; CVSHOPE.com; Throwing up; Puking; Dry heaving; Food poisoning; Episodes; Repeated food poisoning
MeSH Terms: conditions — Familial cyclic vomiting syndrome; Vomiting; Migraine Disorders; Nausea; Abdominal Pain; Foodborne Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- 1mg AZ010 (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: 1mg AZ010
- 3mg AZ010 (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: 3mg AZ-010
- Placebo (Experimental): Single orally-inhaled dose
  Interventions: Combination Product: Staccato Placebo

INTERVENTIONS:
Combination Product: 3mg AZ-010 — Subjects who received a single inhaled dose (3mg)
  Arms: 3mg AZ010
Combination Product: 1mg AZ010 — Subjects who received a single inhaled dose (1mg)
  Arms: 1mg AZ010
Combination Product: Staccato Placebo — Subject who received a single inhaled dose (Staccato Placebo)
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, parallel group, placebo-controlled, efficacy and safety study of adult outpatients diagnosed with CVS and experiencing recurring episodes of stereotypical vomiting.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Safety and Efficacy of Staccato Granisetron (AZ-010) for the Acute Treatment of Moderate to Severe Cyclic Vomiting Syndrome

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females between 18 and 60 years of age, inclusive at the time of signing the informed consent document.
* Diagnosis of cyclic vomiting syndrome (CVS) using the Rome IV diagnostic criteria.
* Otherwise healthy, as determined by the responsible physician, based on a medical evaluation including history, physical examination, vital signs, electrocardiograms (ECGs) and laboratory tests assessed at the screening visit
* Negative urine tests for selected drugs of abuse and alcohol breath test at Screening.

Exclusion Criteria:

* Any significant medical or psychiatric condition that could, in the Investigator's opinion, compromise the subject's safety or interfere with the completion of this protocol.
* Any condition, including the presence of laboratory abnormalities or pulmonary condition, which according to the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
* A diagnosis of any gastrointestinal disorder other than CVS that in the judgement of the Investigator could compromise the subject's safety or interfere with the interpretation of safety or efficacy data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Carter, PhD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (18):
- United States (18):
  - Om Research, Lancaster, California
  - Axis Clinical Trials, Los Angeles, California
  - Precision Research Institute, LLC, San Diego, California
  - University of South Florida, Tampa, Florida
  - Summit Clinical Studies, Athens, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NY Scientific, Brooklyn, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - New Phase Research & Development, LLC, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a multicenter study conducted at 18 sites in the United States. Of these, only 17 sites were activated, and only 15 sites enrolled subjects.
  Study Period: 1 year 5 months Study Start: 05 February 2021 Study End: 26 July 2022 50 patients randomized to each of 3 treatment groups: 1 mg AZ-010, 3 mg AZ-010, or matching Staccato® Placebo Patients were screened at the Research Clinic to determine eligibility for study participation no more than14 days prior to Visit 2.
Pre-assignment Details: Participant eligibility inclusion and exclusion criteria via the following assessments: Medical history (with particular reference to history of vomiting symptoms, CVS diagnosis, typical duration of CVS episode, average # of vomiting/retching events in typical CVS episode, frequency of CVS episodes per year, any triggers for CVS episode, conditions that may cause similar symptoms, treatment history, and current medications, medical history, COVID-19 screening.
Groups:
- 1mg AZ010: Single orally-inhaled dose
  1mg AZ010: Subject will receive a single inhaled dose (1mg)
  single daily dosing up to 5 consecutive days) within 12 weeks after the randomization date.
- 3mg AZ010: Single orally-inhaled dose
  3mg AZ-010: Subject will receive a single inhaled dose (3mg)
  (with single daily dosing up to 5 consecutive days) within 12 weeks after the randomization date.
- Placebo: Single orally-inhaled dose
  Staccato Placebo: Subject will receive a single inhaled dose (Staccato Placebo)
  (with single daily dosing up to 5 consecutive days) within 12 weeks after the randomization date.
Period: Overall Study
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Started | 50 | 51 | 49
Completed | 48 | 48 | 46
Not Completed | 2 | 3 | 3
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Discontinued Prior to Dosing | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- 1mg AZ010: Single orally-inhaled dose
  1mg AZ010: Subject will receive a single inhaled dose (1mg)
- 3mg AZ010: Single orally-inhaled dose
  3mg AZ-010: Subject will receive a single inhaled dose (3mg)
- Placebo: Single orally-inhaled dose
  Staccato Placebo: Subject will receive a single inhaled dose (Staccato Placebo)
- Total: Total of all reporting groups
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (11.95) | 36.0 (12.30) | 36.2 (10.22) | 35.2 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 36 | 104
  Male | 16 | 17 | 13 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 5 | 18
  Not Hispanic or Latino | 41 | 45 | 41 | 127
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 3 | 14
  White | 41 | 45 | 44 | 130
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 168.85 (9.166) | 168.73 (9.729) | 168.81 (7.910) | 168.79 (8.919)
Weight [Mean (Standard Deviation); unit: kg] | 83.28 (24.854) | 78.85 (19.500) | 82.08 (26.443) | 81.38 (23.655)
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 28.979 (7.7236) | 27.529 (6.0793) | 28.238 (7.9544) | 28.244 (7.2635)
Childbearing potential (Yes) [Count of Participants; unit: Participants] | 24 | 29 | 27 | 80
Childbearing potential (No) [Count of Participants; unit: Participants] | 26 | 22 | 22 | 70

OUTCOME MEASURES:

1. Primary Outcome: The Number of Vomiting/Retching Events Reported by Study Participants Following Treatment/Dosing During the Home Treament Period.
Description: The primary efficacy endpoint for this study was the number vomiting/retching events in the two hours following initial treatment. Patients recorded the number of vomiting and retching events that they experienced which occurred 2 hours post dose. Observations occurred at 4 time points: 30 minutes post-dose, 1 hour post-dose, 90 minutes post-dose, and 2 hours post-dose.
  While each treatment group contained 47-49 patients, only 22-35 patients per treatment group (~45-70%) recorded vomiting/retching events at any given time point.
  Safety and tolerability of AZ-010 was assessed by evaluating adverse events, vital signs, 12-lead ECG, clinical laboratory results, and physical examination. Clinically significant deteriorations in physical examination findings (in the opinion of the investigator) are captured and summarized as adverse events.
Time Frame: Within the following timepoints: 30, 60, 90 and 120-minutes post-dose.
Population: Per protocol population (CVS patients between 18 and 60 years of age who experienced at least 3 episodes of recurrent vomiting in the last 12 months and 2 episodes in the last 6 months.
Measure: Mean (Standard Deviation); unit: event
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
event
  Number Vomiting & Retching Events, First Available Efficacy Data, 30 minutes post dose: number analyzed (Participants) | 29 | 35 | 24
  Number Vomiting & Retching Events, First Available Efficacy Data, 30 minutes post dose | 0.69 (1.168) | 1.43 (1.975) | 1.33 (2.239)
  Number Vomiting & Retching Events First Available Efficacy Data, 1 hour post dose: number analyzed (Participants) | 29 | 35 | 24
  Number Vomiting & Retching Events First Available Efficacy Data, 1 hour post dose | 1.48 (2.694) | 2.43 (3.099) | 2.13 (3.180)
  Number Vomiting & Retching Events First Available Efficacy Data, 90 minutes post dose: number analyzed (Participants) | 29 | 34 | 22
  Number Vomiting & Retching Events First Available Efficacy Data, 90 minutes post dose | 2.17 (4.243) | 3.32 (3.906) | 2.59 (4.205)
  Number Vomiting & Retching Events First Available Efficacy Data, 2 hours post dose: number analyzed (Participants) | 29 | 34 | 28
  Number Vomiting & Retching Events First Available Efficacy Data, 2 hours post dose | 3.10 (5.576) | 4.21 (5.279) | 2.61 (4.408)
Statistical Analysis 1: Comparison: 1mg AZ010; Null hypothesis is there was no difference between groups treated with AZ-010 (1 mg or 3 mg) and the placebo group in the mean number of vomiting/retching events in the 2 hours following. treatment. Baseline, body weight, height, body mass index, age as covariates, and the treatment group and study site as factors. All statistical tests were 2-sided with a significance value of ≤ 0.05; Test type: Superiority; p = 0.7024, ANOVA
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority — Null hypothesis is there was no difference between groups treated with AZ-010 (1 mg or 3 mg) and the placebo group in the mean number of vomiting/retching events in the 2 hours following. treatment. Baseline, body weight, height, body mass index, age as covariates, and the treatment group and study site as factors. Patients summarized by actual treatment received. Formal statistical tests (ANOVA, when performed) were 2-sided t-tests with a significance value of 0.05; p = 0.2051, ANOVA

2. Secondary Outcome: Anxiety/Panic Visual Analog Scale (VAS) Score
Description: Assessment of anxiety/panic at 2, 6, 12, and 24 hours following treatment. The assessment of anxiety/panic Visual Analog Scale (VAS) score whereby 0 = no anxiety/panic and 100 = worst possible anxiety/panic 0-100; 0 = no anxiety/panic and 100 = worst possible anxiety/panic).
  Participants were asked to rate their anxiety/panic on scale of 0-100 at each time point. The higher the number, the more intense the symptom.
Time Frame: 24 hours after treatment dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
score on a scale
  Anxiety/Panic VAS Score, 2 hour, post-dose: number analyzed (Participants) | 23 | 26 | 25
  Anxiety/Panic VAS Score, 2 hour, post-dose | 51.30 (34.907) | 52.08 (35.020) | 47.72 (32.849)
  Anxiety/Panic VAS Score, 6 hour, post-dose: number analyzed (Participants) | 8 | 8 | 7
  Anxiety/Panic VAS Score, 6 hour, post-dose | 48.25 (17.343) | 64.00 (35.071) | 51.29 (20.605)
  Anxiety/Panic VAS Score, 12 hour, post-dose: number analyzed (Participants) | 3 | 13 | 4
  Anxiety/Panic VAS Score, 12 hour, post-dose | 31.00 (28.827) | 51.15 (31.947) | 64.00 (26.533)
  Anxiety/Panic VAS Score, 24 hour, post-dose: number analyzed (Participants) | 5 | 8 | 4
  Anxiety/Panic VAS Score, 24 hour, post-dose | 18.00 (19.378) | 37.88 (31.439) | 62.25 (30.478)
Statistical Analysis 1: Comparison: 1mg AZ010; Participants were asked to rate their anxiety/panic on scale of 0-100 at each time point. The higher the number, the more intense the symptom; Test type: Superiority; p = 0.0504, Mixed Models Analysis
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority — Participants were asked to rate their anxiety/panic on scale of 0-100 at each time point. The higher the number, the more intense the symptom; p = 0.8246, Mixed Models Analysis

3. Secondary Outcome: Prior Episode Questionnaire
Description: The duration of the CVS episode at 24 hours in relation to their typical CVS episodes (Prior Episode Questionnaire) and the intensity of the CVS episode at 24 hours in relation to their typical CVS episodes. A 3-point scale was used. The questions were prompted approximately 24 hours after each dose of study medication was administered.
  Duration: (Score definition: 1 = shorter duration than typical previous episode; 2 = same duration as typical previous episode; 3 = longer duration than typical previous episode) Intensity: (Score definition: 1 = less intense than typical previous episode; 2 = same intensity as typical previous episode; 3 = more intense than typical previous episode)
Time Frame: 24 hours after each dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
score on a scale
  Prior Episode Questionnaire, 24 Hours Post-Dose, Duration Of Current Episode: number analyzed (Participants) | 24 | 22 | 21
  Prior Episode Questionnaire, 24 Hours Post-Dose, Duration Of Current Episode | 1.46 (0.658) | 1.27 (0.550) | 1.52 (0.680)
  Prior Episode Questionnaire, 24 Hours Post-Dose, Intensity Of Current Episode: number analyzed (Participants) | 24 | 22 | 21
  Prior Episode Questionnaire, 24 Hours Post-Dose, Intensity Of Current Episode | 1.58 (0.654) | 1.55 (0.671) | 1.43 (0.598)
Statistical Analysis 1: Comparison: 1mg AZ010; Test type: Superiority; p = 0.8299, Mixed Models Analysis — Prior Episode Duration 1mg AZ-010
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.2346, Mixed Models Analysis — Prior Episode Duration 3 mg AZ-010
Statistical Analysis 3: Comparison: 1mg AZ010; Test type: Superiority; p = 0.3997, Mixed Models Analysis — Prior Episode intensity 1mg AZ-010
Statistical Analysis 4: Comparison: 3mg AZ010; Test type: Superiority; p = 0.3997, Mixed Models Analysis — Prior Episode intensity 3mg AZ-010

4. Secondary Outcome: Rescue Medication Use Within 1 Day of Dose
Description: The percentage of patients who used rescue medication within the first day of treatment; patients confirming the individual had used some sort of rescue medication.
Time Frame: 24 hours post dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
Participants
  Percentage of patients confirming "Yes" response to rescue medication use, 2 hours post dose: number analyzed (Participants) | 31 | 36 | 33
  Percentage of patients confirming "Yes" response to rescue medication use, 2 hours post dose | 3 | 2 | 1
  Percentage of patients confirming "Yes" response to rescue medication use, 24 hours post dose | 9 | 11 | 6
Statistical Analysis 1: Comparison: 1mg AZ010; Test type: Superiority; p = 0.3847, Mantel Haenszel
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.1785, Mantel Haenszel

5. Secondary Outcome: Health Care Provider Visits; Visit to Urgent Care, Emergency Department, or Physician's Office
Description: Health Care Provider Visits; Visit to Urgent Care, Emergency Department, or Physician's Office for care within the first day following dosing for a CVS episode.
Time Frame: Within Day 1 after dosing
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
Participants
  Patients requiring healthcare provider visit within 24 hours post dose of CVS episode. | 2 | 0 | 0
  Patients not requiring healthcare provider visit within 24 hours post dose of CVS episode. | 45 | 49 | 44
Statistical Analysis 1: Comparison: 1mg AZ010; Test type: Superiority; p = 0.9732, Mantel Haenszel
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.1471, Mantel Haenszel

6. Secondary Outcome: Rhodes Index of Nausea, Vomiting, and Retching (RINVR)
Description: The Rhodes Index of nausea, vomiting, and retching (RINVR) at 6, 12, and 24 hours following treatment. The Rhodes Index of nausea, vomiting, and retching (RINVR) is designed to assess the degree of nausea distress and vomiting distress in patients. It is composed of 8 questions, and each question has 5 choices. The 5 choices for each individual question are scores from 0 to 4, with 0 being the lowest level without any symptoms related to nausea/vomiting/retching and 4 being the highest level. Individual question scores can be tracked over time, or a composite score with a total scoring range of 0 to 32 can be formed by adding the individual scores of the symptom occurrence and degree of discomfort questions together. Composite scores classified as follows: 0: no symptoms, 1-8: mild, 9-16: moderate, 17-24: great, 25-32: severe. This scale was adapted for the ePD, and patients were prompted to answer the questions according to the Schedule of Events.
Time Frame: Within 24 hours following treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
score on a scale
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 6 hour, post-dose: number analyzed (Participants) | 25 | 26 | 28
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 6 hour, post-dose | 11.20 (7.741) | 11.85 (7.893) | 11.79 (7.695)
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 12 hour, post-dose: number analyzed (Participants) | 23 | 31 | 21
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 12 hour, post-dose | 6.57 (7.710) | 10.45 (9.237) | 7.81 (8.274)
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 24 hour, post-dose: number analyzed (Participants) | 25 | 23 | 25
  Rhodes Index of Nausea, Vomiting and Retching (RINVR) Composite Score, 24 hour, post-dose | 6.76 (7.096) | 8.87 (8.471) | 7.92 (8.057)
Statistical Analysis 1: Comparison: 1mg AZ010; The RINVR is an 8-part questionnaire with each item scored from 0-4, for a total scoring range of 0-32. A lower score indicates less distress related to nausea, vomiting, and retching. The data shown is collected within the first 24 hours after the first at-home dose; Test type: Superiority; p = 0.1337, ANOVA
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.7224, ANOVA

7. Secondary Outcome: Abdominal Pain, Visual Analog Scale (VAS) Score
Description: The patient was asked the abdominal pain in relation to their last vomiting/retching episode, whereby 0 = no pain and 100 = worst possible pain at timepoints 2, 6, 12 and 24 hours post-dose
Time Frame: Up to 24 hours post dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
units on a scale
  Abdominal Pain VAS Score,2 hour, post-dose: number analyzed (Participants) | 23 | 26 | 25
  Abdominal Pain VAS Score,2 hour, post-dose | 45.48 (27.318) | 53.04 (32.227) | 51.60 (29.390)
  Abdominal Pain VAS Score,6 hour, post-dose: number analyzed (Participants) | 8 | 8 | 7
  Abdominal Pain VAS Score,6 hour, post-dose | 51.50 (17.849) | 47.25 (33.970) | 32.57 (22.846)
  Abdominal Pain VAS Score,12 hour, post-dose: number analyzed (Participants) | 3 | 13 | 4
  Abdominal Pain VAS Score,12 hour, post-dose | 36.67 (7.024) | 51.38 (33.393) | 61.25 (30.489)
  Abdominal Pain VAS Score, 24 hour, post-dose: number analyzed (Participants) | 5 | 8 | 4
  Abdominal Pain VAS Score, 24 hour, post-dose | 32.60 (17.771) | 43.88 (38.264) | 66.25 (11.354)
Statistical Analysis 1: Comparison: 1mg AZ010; Participants were asked to rate their abdominal pain, nausea, and anxiety/panic on scale of 0-100 at each time point. The higher the number, the more intense the symptom; Test type: Superiority; p = 0.0504, Mixed Models Analysis
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.8246, Mixed Models Analysis

8. Secondary Outcome: Intensity of Vomiting/Retching Attack
Description: The Intensity of Attack scale assessed the severity of the last vomiting/retching episode at 2, 6, 12, and 24 hours post dose.
  Intensity of attack is evaluated on a scale of 1-4 (1=Mild, 2=Moderate, 3=Severe, 4=Excruciating).
Time Frame: Within 24 hours post dose.
Population: Per protocol population (CVS patients between 18 and 60 years of age who reported intensity of vomiting attack.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
Number analyzed (Participants) | 47 | 49 | 48
units on a scale
  Intensity of Attack Scale (Efficacy Population) 2 hours post-dose: number analyzed (Participants) | 7 | 6 | 4
  Intensity of Attack Scale (Efficacy Population) 2 hours post-dose | 2.29 (0.488) | 3.00 (0.894) | 2.25 (0.957)
  Intensity of Attack Scale (Efficacy Population) 6 hour, post-dose: number analyzed (Participants) | 7 | 7 | 7
  Intensity of Attack Scale (Efficacy Population) 6 hour, post-dose | 1.86 (0.690) | 2.29 (0.756) | 1.57 (0.787)
  Intensity of Attack Scale (Efficacy Population) 12 hour, post-dose: number analyzed (Participants) | 3 | 13 | 4
  Intensity of Attack Scale (Efficacy Population) 12 hour, post-dose | 1.33 (0.577) | 2.31 (0.947) | 1.75 (0.957)
  Intensity of Attack Scale (Efficacy Population) 24 hour, post-dose: number analyzed (Participants) | 5 | 8 | 4
  Intensity of Attack Scale (Efficacy Population) 24 hour, post-dose | 2.20 (0.837) | 2.38 (0.916) | 2.25 (0.957)
Statistical Analysis 1: Comparison: 1mg AZ010; Test type: Superiority; p = 0.9664, Mixed Models Analysis
Statistical Analysis 2: Comparison: 3mg AZ010; Test type: Superiority; p = 0.7919, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: up to 30 days after the last dose
Arm/Group | 1mg AZ010 | 3mg AZ010 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 3/50 | 3/51 | 3/49
Other Adverse Events (participants affected / at risk) | 28/50 | 40/51 | 44/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1mg AZ010 (N=50) | 3mg AZ010 (N=51) | Placebo (N=49)
CVS, Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — 3 mg AZ-010
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Placebo
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1mg AZ010 (N=50) | 3mg AZ010 (N=51) | Placebo (N=49)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (13) | 2 (2) — 1mg, 3mg, placebo AZ010
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) — 1mg, 3mg, placebo AZ010
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) — 1mg, 3mg, placebo AZ010
Stomach pain (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1) — 3mg, placebo AZ010
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — 3mg AZ010
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Bloated Feeling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Erosive esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Gas pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Gastroesohageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Hematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Pain abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Vomited (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 4 (4) — 1mg, placebo AZ010
Burning sensation (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) — 3mg AZ010
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) — 1mg, 3mg, placebo AZ010
Acute diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Acute pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Yeast infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) — 1mg, 3mg placebo AZ010
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) — 3mg, placebo AZ010
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3) — placebo AZ010
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) — 1mg, placebo AZ010
Depersonalization (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0) — 3mg AZ010
Difficulty sleeping (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) — 1mg, 3mg AZ010
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — 3mg, placebo AZ010
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) — 3mg AZ010
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) — 3mg, placebo AZ010
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Poikilothermia (General disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Tiredness (General disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Generalized muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — 1mg, placebo AZ010
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Weakness in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Pale skin (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Endoscopic retrograde cholangiopancreatography (Investigations) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Lactate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
QT interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
ST segment depressed (Investigations) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010
Transaminitis (Investigations) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) — 3mg AZ010
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Left anterior fascicular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Palpitations (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) — 3mg AZ010
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Gallstones (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Knee injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Car sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) — placebo AZ010
Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — 3mg AZ010
Menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — placebo AZ010
Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — 1mg AZ010

LIMITATIONS AND CAVEATS:
The complexity of data collection interface/instructions and patient impairment while experiencing severe CVS episodes may likely have led to the high incidence of missing data with impaired patients missing data collection timepoints. A simplified data collection interface, clear instructions, and potentially collection of fewer overall parameters may make it easier for patients in future studies to record complete study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alexza Pharmaceuticals has full ownership of the data collected as part of the study. The results of this study may be published in a medical publication, journal, or another public dissemination, presented at a medical conference or used for teaching purposes. This study and its results may be submitted for inclusion in all appropriate health authority study registries, as well as publication on health authority study registry websites, as required by local health authority regulations.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT04645953/Prot_SAP_000.pdf